CLINICAL TRIAL: NCT00071149
Title: Consistency of Traditional Chinese Medicine Rheumatoid Arthritis Diagnosis and Herbal Prescriptions
Brief Title: Consistency of Traditional Chinese Medicine Diagnoses and Herbal Prescriptions for Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R21AT000590-01 (NIH)
Record Dates: First submitted 2003-10-14; First posted 2003-10-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; TCM; Diagnosis; Traditional Chinese Medicine; Complementary Therapies
MeSH Terms: conditions — Arthritis, Rheumatoid; Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Practitioners of Traditional Chinese Medicine (TCM) make diagnoses based solely on clinical symptoms. This study will evaluate whether TCM practitioners make diagnoses consistently.

DETAILED DESCRIPTION:
TCM is one of the oldest and most widely-used indigenous medical systems in the world. It is difficult to effectively practice or evaluate TCM outside of its core framework, which includes a diagnostic system that is more conceptual and less technologically driven than that of conventional medicine. TCM diagnosis relies entirely on clinical symptoms and signs that are discerned by the practitioner. The establishment of diagnostic and prescriptive consistency is crucial for efficacy studies involving individualized treatments within the TCM framework. This study will examine the consistency of TCM diagnoses and herbal prescriptions under controlled conditions.

Rheumatoid arthritis (RA) patients will be individually evaluated by three TCM practitioners; the diagnostic and prescriptive behaviors of the practitioners will be recorded and analyzed to determine: 1) the extent to which two or more TCM practitioners assign comparable TCM diagnoses to the same RA patients; 2) the extent to which two or more TCM practitioners prescribe comparable herbal formulas to the same RA patients; and 3) the extent to which TCM diagnoses are related to conventional clinical assessments and biomedical tests of RA. Variables that cause inconsistency will be identified and analyzed.

ELIGIBILITY:
Inclusion Criteria

* Rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-11; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Grant G Zhang, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States